CLINICAL TRIAL: NCT06283407
Title: Comparative Analysis of the Musculoskeletal Health of General Population in Poland and Spain: a Cross-sectional Study Using the International Classification of Functioning, Disability and Health for Chronic Musculoskeletal Conditions
Brief Title: ICF-based Comparison on Musculoskeletal Health in Poland and Spain
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rzeszow (Other)
Collaborators: Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Agnieszka Wiśniowska-Szurlej, PhD, University of Rzeszow
Other Study IDs: ICF
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: International Classification of Functioning, Disability and Health; Musculoskeletal Diseases;; Disability Evaluation; Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Poland: People with musculoskeletal conditions from the general population in Poland
  Interventions: Other: ICF-based cross-country comparative analysis
- Spain: People with musculoskeletal conditions from the general population in Spain
  Interventions: Other: ICF-based cross-country comparative analysis

INTERVENTIONS:
Other: ICF-based cross-country comparative analysis — ICF-based cross-country comparative analysis

SUMMARY:
Musculoskeletal conditions are a major cause of disability worldwide. These conditions are often associated with chronicity, which is a challenge for healthcare systems to address. Health care must be person-centred and take into account the individual perspective from which the disease is experienced. The lived experience of health conditions depends to a large extent on contextual factors. Comparison between different contexts helps to identify which aspects are most relevant in the experience of the disease. The International Classification of Functioning, Disability and Health (ICF) provides a unified language that allows such comparisons to be made. The aim of this study is to identify differences in musculoskeletal health between the Polish and Spanish populations using the ICF as a frame of reference.

DETAILED DESCRIPTION:
Musculoskeletal conditions are a major cause of disability worldwide. These conditions are often associated with chronicity, which is a challenge for healthcare systems to address. Health care must be person-centred and take into account the individual perspective from which the disease is experienced. The lived experience of health conditions depends to a large extent on contextual factors.

The ICF is the framework proposed by the World Health Organization to describe the organic changes caused by a condition and the modulating effect of contextual factors on the resulting disability. The ICF core sets are tools that facilitate the use of this classification in clinical practice. The ICF core sets have been developed for a wide range of health conditions, but there has traditionally been a lack of validation studies. In recent years, studies have been developed using ICF core sets for musculoskeletal conditions in different populations. In particular, the musculoskeletal health of the Polish and Spanish populations has been assessed using the brief ICF core set for post-acute musculoskeletal conditions. This availability of data allows comparisons to be made of the health status of these populations using the ICF as a frame of reference. This possibility of using ICF for this purpose is unknown in the scientific literature and could contribute to the identification of the aspects that are most relevant in the experience of the health condition.

The aim of this study is to identify differences in musculoskeletal health between the Polish and Spanish populations using the ICF as a frame of reference. The development of this study also has the aim of providing the methodological basis for the development of transnational comparisons on the basis of the ICF.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years,
* diagnosed musculoskeletal disorder according to ICD-10,
* normal cognitive status to perform reliable study (The Abbreviated Mental Test Score >6),
* informed and voluntary consent to participate in the study,
* sufficient knowledge of the Spanish or Polish language.

Exclusion Criteria:

* mental disorders - depression or personality disorders confirmed by a medical diagnosis,
* referral for a non-musculoskeletal problem,
* referral from hospital services.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with musculoskeletal conditions from the general population in Poland and Spain will be the potential participants in this study.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-06-03 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
Brief International Classification of Functioning, Disability and Health (ICF) core set for post-acute musculoskeletal conditions | 2024-01/2024-07
  The core set of codes cover categories, including Body Functions, Activities and Participation and Environment Factors. All codes from each category are quantitatively assessed with qualifiers using the same scale denoting the severity of the problem or the magnitude of the impairment on a scale of 0 to 4 (xxx.0 NO problem; xxx.1 MILD problem; xxx.2 MODERATE problem; xxx.3 SEVERE problem; xxx.4 COMPLETE problem; xxx.8 not specified and xxx.9 not applicable).

SECONDARY OUTCOMES:
Sociodemographic data of the sample (nationality, age, sex, education level, work status, number of comorbidities) | 2024-01/2024-07

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Wiśniowska-Szurlej, PhD, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszow, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisniowska-Szurlej A, Sozanska A, Barrio SJ, Sozanski B, Ceballos-Laita L, Hernandez-Lazaro H. ICF based comparison of musculoskeletal health in regions of Poland and Spain. Sci Rep. 2024 Nov 12;14(1):27671. doi: 10.1038/s41598-024-77450-2. PMID 39532934